CLINICAL TRIAL: NCT04686084
Title: A Clinical Trial to Evaluate the Effectiveness and Safety of Dual Energy Cone-Beam Computed Tomography (DE-CBCT) Imaging for Quantitative Measurement of Jaw Bone Density
Brief Title: Dual Energy Cone-Beam Computed Tomography (DE-CBCT) Assessment of Jaw Bone Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Sanjay Mallya, BDS, MDS, PhD, Associate Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-001768
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Dental Diseases
Keywords: cone beam computed tomography, dual-energy CT
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CT scan (Experimental): CT scan (MDCT, standard of care) and DE-CBCT (Investigational)
  Interventions: Device: Dual-energy computed tomography scan

INTERVENTIONS:
Device: Dual-energy computed tomography scan — Diagnostic CT scan

SUMMARY:
Current radiologic imaging modalities used in dentistry provide information on the morphology of the hard tissues. Additional information on the density of bone has practical relevance, for example, in dental implant treatment planning, where local bone quality is a known strong predictor of successful implant osseointegration. The Dual-Energy Cone Beam Computed Tomography (DE-CBCT) device is designed to overcome limitations of traditional imaging and will provide assessment of jaw bone density in additional to morphological information.

This clinical trial will examine the application of DE-CBCT to assess jaw bone density and compare Hounsfield units (HU) values with multidetector CT, an established standard for assessing BD.

DETAILED DESCRIPTION:
This is a single center, open-label trial, designed to enroll 24 patients. Both, the researcher and the subject know the treatment the participant is receiving.

To evaluate the effectiveness and safety of DE-CBCT to evaluate jaw bone density and compare HU values with those of multidetector CT, an established standard for assessing BD.

The study is based on two visits (VISIT 1 and VISIT 2) • DAY 0 (enrollment): Subject is queried for inclusion/exclusion criteria and informed about the study. If he/she agrees to participate, inclusion/exclusion criteria and informed consent will be documented. An imaging stent, which bears radiopaque markers, will be also created for each patient.

• VISIT 1: Inclusion/exclusion criteria will be reconfirmed and the DE-CBCT imaging will be completed.

• VISIT 2 (no more than 30 days since the enrollment): Inclusion/exclusion criteria will be reconfirmed and MDCT imaging completed.

- Depending on availability of scheduling on MDCT unit, Visit 2 may occur on the same day as Visit 1.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need x-ray imaging for dental treatment planning and/or diagnosis
2. Males or females aged older than 21
3. Can follow instructions to be positioned into the CT scanner
4. Can remain physically immobile during the CT scan acquisition
5. Voluntarily sign and date the informed consent

Exclusion Criteria:

1. Pregnancy
2. Patients who are unable to comprehend the risks of the study to provide informed consent
3. Extensive dental restorations, maxillofacial prosthesis, or orthopedic hardware that likely may cause artifacts and degrade quality, as determined by the study radiologists

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay M Mallya, BDS,MDS,PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA School of Dentistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CT Scans: MDCT scan (Standard of care procedure, 1 scan) DE-CBCT (Investigational procedure, 1 scan)
Period: Overall Study
Arm/Group | CT Scans
Started | 26
Completed | 25
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | CT Scan
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Bone Density Assessment
Description: Bone density (g/cc) in a region of interest measured by the OnDemand software
Time Frame: 30 days
Population: Patients imaged with MDCT and DE-CBCT
Measure: Mean (Standard Deviation); unit: g/cc
Groups:
- CT Scan: CT scan (MDCT, standard of care)
- DE-CBCT Scan (Investigational): Patients imaged with the dual energy CBCT scan
Arm/Group | CT Scan | DE-CBCT Scan (Investigational)
Number analyzed (Participants) | 25 | 25
g/cc | 0.48 (0.31) | 0.46 (0.36)
Statistical Analysis 1: Comparison: CT Scan vs DE-CBCT Scan (Investigational); Test type: Other — Bland-Altman analysis; Median Difference (Final Values) = 0.04

ADVERSE EVENTS:
Time Frame: At time of study scan, up to 30 days
Arm/Group | CT Scan
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04686084/Prot_SAP_000.pdf